CLINICAL TRIAL: NCT00308113
Title: PITT0503: Clinical Trial of Coenzyme Q10 and Prednisone in Duchenne Muscular Dystrophy
Brief Title: CoQ10 and Prednisone in Non-Ambulatory DMD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: New enrollment has been suspended, currently following previously enrolled participants
Sponsor: Cooperative International Neuromuscular Research Group (Network)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PITT0503
Record Dates: First submitted 2006-03-27; First posted 2006-03-29 (Estimated); Results first posted 2013-10-11 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-10

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Muscular dystrophy; Duchenne; CoQ10; prednisone
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies | interventions — Prednisone; coenzyme Q10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): CoenzymeQ10 taken once a day each morning by mouth.
  Interventions: Dietary Supplement: Coenzyme Q10
- 2 (Active Comparator): Prednisone taken once a day each morning by mouth
  Interventions: Drug: Prednisone
- 3 (Active Comparator): CoenzymeQ10 and prednisone each taken once a day in the morning by mouth.
  Interventions: Drug: Prednisone; Dietary Supplement: Coenzyme Q10
- 4 (No Intervention): Enhanced standard of care.

INTERVENTIONS:
Drug: Prednisone — Prednisone 0/75 mg/kg/day.
  Arms: 2; 3
Dietary Supplement: Coenzyme Q10 — serum levels of greater or equal to 2.5 micrograms/mL.
  Other Names: CoQ10
  Arms: 1; 3

SUMMARY:
This study will help determine if CoQ10 and prednisone, alone and as a combination decrease the decline in cardiopulmonary and skeletal muscle function that occurs in the wheelchair confined phase of DMD. Participants who are enrolled in this study should not have taken any corticosteroids within the last six months. This is a 13-month, prospective, randomized study comparing a daily prednisone arm (0.75mg/kg/day), a CoQ10 arm (serum of greater than 2.5 ug/mL) and a combination arm (prednisone and CoQ10) with an enhanced standard of care arm in wheelchair confined males age 10 to 18 years with an established DMD diagnosis.

DETAILED DESCRIPTION:
Duchenne muscular dystrophy (DMD) is the most common form of muscular dystrophy affecting 1:3500 male births worldwide. Despite an increase in our understanding of the disorder since the discovery and characterization of the causative gene and its product dystrophin in 1987, current therapeutic management remains largely supportive. Improvement in the treatment of DMD will depend upon the development of better therapies. Affected boys become symptomatic at 3 to 5 years of age with proximal leg weakness that impairs mobility, ability to get up from a squat, and precludes a normal ability to run. By 8 years of age, some affected boys begin to lose the ability to walk and resort to a wheelchair for mobility. This shift from the ambulant to non-ambulant phase occurs in all boys with a diagnosis of DMD by age 12 years. In this study, participants will be randomized into groups after being screened to determine eligibility. Participants will then be followed for a 12-month investigation period.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-18 years
* Non-ambulatory (primary mode of transportation is via wheelchair for 3 years or less)
* Confirmed DMD diagnosis
* Steroid-naive for the 6 months prior to screening
* Stable dose of b-blocker or ACE inhibitor medication for the 6 months prior to screening, if taking either of these medications
* Ability to provide reproducible repeat QMT grip score within 15% of first assessment score
* Has not participated in other therapeutic research protocol within the last 6 months prior to screening
* Ability to swallow tablets

Exclusion Criteria:

* Failure to achieve one or more of the diagnostic inclusion criteria cited above
* Symptomatic DMD carrier
* Use of carnitine, other amino acids, creatine, glutamine, CoQ10 or any herbal medicines (this would not include herbal teas unless they are consumed daily with intended medicinal effect) within the last 3 months
* History of significant concomitant illness or significant impairment of renal or hepatic function, or other contraindication to steroid therapy
* Positive PPD
* No prior exposure to chickenpox and no immunization against chicken pox
* Baseline serum CoQ10 level of 5.0mg/ml or greater

Ages: 10 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2007-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula R Clemens, M.D., Study Chair — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in April 2007 at two participating centers of the Cooperative International Neuromuscular Research Group (CINRG): University of Pittsburgh and University of Puerto Rico. Enrollment closed in December 2008 by the CINRG Data and Safety Monitoring Board (DSMB) due to changes in standard of care.
Groups:
- Coenzyme Q10 Alone: CoenzymeQ10 taken once a day each morning by mouth.
  Coenzyme Q10 : serum levels of greater or equal to 2.5 micrograms/mL.
- Prednisone Alone: Prednisone taken once a day each morning by mouth
  Prednisone : Prednisone 0/75 mg/kg/day.
- Coenzyme Q10 and Prednisone: CoenzymeQ10 and prednisone each taken once a day in the morning by mouth.
  Coenzyme Q10 : serum levels of greater or equal to 2.5 micrograms/mL.
  Prednisone : Prednisone 0/75 mg/kg/day.
- Enhanced Standard of Care: Enhanced standard of care.
Period: Overall Study
Arm/Group | Coenzyme Q10 Alone | Prednisone Alone | Coenzyme Q10 and Prednisone | Enhanced Standard of Care
Started | 0 | 0 | 1 | 2
Completed | 0 | 0 | 1 | 1
Not Completed | 0 | 0 | 0 | 1
Not completed — Protocol closure | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Coenzyme Q10 Alone | Prednisone Alone | Coenzyme Q10 and Prednisone | Enhanced Standard of Care | Total
Number analyzed (Participants) | 0 | 0 | 1 | 2 | 3
Age, Customized [Number; unit: participants]
  10-18 years |  |  | 1 | 2 | 3
Gender [Number; unit: participants]
  Female |  |  | 0 | 0 | 0
  Male |  |  | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: One Year Change of Left Ventricular Mean Systolic Wall Stress/Rate-corrected Velocity of Fiber Shortening Relation.
Description: Comparing change from baseline of mean systolic wall stress and rate-corrected mean velocity of circumferential shortening in the three treatment groups relative to the enhanced standard of care group and relative to each other at one year. The values are obtained via an echocardiogram read locally at each site.
Time Frame: 12 months
Population: No analysis was performed as only 1 out of 3 participants completed all echocardiogram measurements before the protocol was closed.
Arm/Group | Coenzyme Q10 Alone | Prednisone Alone | Coenzyme Q10 and Prednisone | Enhanced Standard of Care
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: One Year Change in Pulmonary Function (Forced Expiratory Volume, FEV1 and Forced Vital Capacity, FVC)
Description: Comparing change from baseline levels in pulmonary function (FEV1 and FVC) in the three treatment groups relative to the enhanced standard of care group and relative to each other at one year.
Time Frame: 12 months
Population: No analysis was performed as only 1 out of 3 participants completed all the pulmonary function measurements before the protocol was closed.
Arm/Group | Coenzyme Q10 Alone | Prednisone Alone | Coenzyme Q10 and Prednisone | Enhanced Standard of Care
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Compare Side Effect Profiles of the Three Study Groups
Description: To compare side effect profiles of the three regimens to the enhanced standard of care group, to include height, weight, weight/height ratio, body mass index, cataract formation, blood glucose, blood pressure, and behavioral changes.
Time Frame: 12 months
Population: No analysis was performed as the study was closed with N=3 out of 120 and side effects profile between groups could not be analyzed.
Arm/Group | Coenzyme Q10 Alone | Prednisone Alone | Coenzyme Q10 and Prednisone | Enhanced Standard of Care
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Coenzyme Q10 Alone | Prednisone Alone | Coenzyme Q10 and Prednisone | Enhanced Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 1/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 1/1 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Coenzyme Q10 Alone (N=0) | Prednisone Alone (N=0) | Coenzyme Q10 and Prednisone (N=1) | Enhanced Standard of Care (N=2)
Tonsilectomy (Surgical and medical procedures) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Coenzyme Q10 Alone (N=0) | Prednisone Alone (N=0) | Coenzyme Q10 and Prednisone (N=1) | Enhanced Standard of Care (N=2)
Limb edema (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Cardiac arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Upper airway infection (Infections and infestations) | 0 | 0 | 1 | 0
Mood alteration and agitation (General disorders) | 0 | 0 | 1 | 0
Gastrointestinal Virus (Gastrointestinal disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
In December 2007 the CINRG Data Safety and Monitoring Board (DSMB) met and recommended to close the study as the AAN had released practice parameters recommending that all patients with DMD should be offered treatment with corticosteroids.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No